CLINICAL TRIAL: NCT05530187
Title: Testing a Model of Care Based on Electronic Patient Reported Outcome Monitoring for Patients With Cancer Under Immune-checkpoint Blockade: A Phase II Study (IePRO Study)
Brief Title: ePRO-based Model of Care to Manage and Monitoring Symptoms of Cancer Patients Treated With Immune Checkpoint Inhibitors
Acronym: IePRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manuela Eicher (Other)
Responsible Party: Sponsor-Investigator, Manuela Eicher, Associate Professor and Director at Faculty of Biology and Medicine, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IePRO
Record Dates: First submitted 2022-08-31; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Patient Reported Outcome Measures; Patient Safety
Keywords: Patient-reported outcomes; Model of care; Remote symptom monitoring; Immune-related adverse events; PRO; IrAE

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental)
  Interventions: Device: Electronic Patient-reported Outcomes-based Model of Care

INTERVENTIONS:
Device: Electronic Patient-reported Outcomes-based Model of Care — Patients in the intervention arm of this study will report symptoms weekly through an electronic symptom questionnaire. For the first 3 months of the 6 month intervention, they will reassess the reported symptoms daily. A team of oncology nurses will contact patients by telephone if they declare a new or worsening symptom. The nurses will use a triage algorithm to identify patient needs (self-care, remote follow-up or in-person assessment).
  Arms: Intervention

SUMMARY:
Immune checkpoint inhibitors (ICIs) can cause immune-related adverse events (IrAEs) throughout and beyond treatment duration. These IrAEs can be varied and difficult to predict, as they can involve almost any organ, regardless of where the primary tumor is located. Treatment modality and individual characteristics appear to influence the frequency and severity of these events, which can become serious without proper monitoring and timely intervention.

Generally, patient visits are scheduled at the same intervals in which patients receive treatment, once every two to four weeks. In these large intervals, patients can be surprised by IrAEs without a close schedule visit to their oncology physician. Not only this may negatively influence their overall well-being, their perceived self-efficacy to manage their own condition and their health-related quality of life may be affected as well.

Using patient-reported outcomes (PROs) to monitor patient symptoms has become incredibly valuable in describing treatment toxicity, including that of ICIs. PROs are a self-report of the patient's own perceptions of their health status. Using their own words, or by replying to questionnaires, patients can convey symptoms and how these affect their daily life and quality of life.

Questionnaires are an example of a PRO measure (PROM), which have increasingly been provided electronically (resulting in electronic PROs or ePROs). The ubiquity of connected electronic devices has enabled long-distance monitoring of symptoms through electronic questionnaires. In patients treated with chemotherapy, studies have shown that using this method to collect symptom data can enable healthcare providers to help patients manage their symptoms remotely. This allows patients to receive timely support from home, that could help prevent serious complications that could entail visits to the emergency department, unscheduled hospitalizations and treatment interruptions.

The IePRO study's aim is to test a model of care that uses electronic questionnaires to monitor symptoms that could be related to the use of ICIs. Patients would reply to these questionnaires at least once a week using an electronic web application (on their phone or computer). A team of oncology nurses reviews their replies and calls patients when new symptoms appear or when they worsen. Using a standard triage algorithm, the nurses guide patients on how to proceed: if they should stay home and follow self-care advice, if they should have a second call within the next 24 hours to follow-up on their symptoms, or if they should come to the hospital for an in-person assessment as soon as possible.

In this study, it is hypothesized that this model of care could lead to an earlier detection of IrAEs, as well as their improved management by reducing the number of high-severity IrAEs, the number of unscheduled emergency admissions and hospitalizations, as well as decreasing the number of treatment interruptions and of immunosuppressive treatments used to treat IrAEs.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or older
* Patients diagnosed with cancer
* Patients starting or re-starting systemic ICI therapy treatments (adjuvant, neo-adjuvant, metastatic)
* Informed Consent as documented by signature

Exclusion Criteria:

* Patients that self-declare not being able to use an ePRO application and complete a questionnaire in French.
* Patients with any psychological, familial or sociological condition and linguistic limitation potentially hampering compliance with the study protocol requirements and/or follow-up procedures. These conditions will be discussed between the recruiting oncologist and the patient before trial entry.
* Patients that are re-starting ICI therapy, but that have previously participated in this intervention.
* Patients with a cognitive impairment, as declared in the patient record
* Patients participating in other interventional clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-11-02 (Estimated); Study Completion 2023-11-02 (Estimated)

PRIMARY OUTCOMES:
IrAE time-to-detection | Through study completion, an average of 6 months
  The primary outcome is the difference (in days) between the symptom onset date and the date when it was detected by the oncology team.

SECONDARY OUTCOMES:
Number of symptomatic IrAEs experienced by patients | Up to 6 months
  Number, type and grade of diagnosed Symptomatic IrAEs.
Number of self-reported symptoms | Up to 6 months
  Type and number of self-reported PRO-CTCAE items.
Symptom-to-treatment interval | Up to 6 months
  Time (in days) between symptom onset and the first pharmacological intervention for the symptomatic IrAE.
IrAE treatments | Up to 6 months
  Number and type of documented pharmacological interventions to manage IrAEs.
Maximum IrAE grade | Up to 6 months
  Highest recorded IrAE grade according to the CTCAE version 5.0
Health-related Quality of Life score measured with the FACT-G questionnaire | Up to 6 months
  Change from baseline in health-related quality of life (weekly and at 6 months)
Self-efficacy score as measured with the PROMIS Self-Efficacy for Managing Symptoms short form 8a questionnaire | Up to 6 months
  Change from baseline in perceived self-efficacy to manage symptoms (weekly and at 6 months)
Overall survival | Up to 6 months
  Overall survival at 6 months.
Triage process | Up to 6 months
  Type and amount of IrAE management actions/instructions issued by triage nurses, per resulting alerts (green, amber and red alerts).

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud
  - Hôpitaux Universitaires de Genève, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopes AMDS, Giacomini S, Ulahannan A, Darnac C, Bugeia S, Gutknecht G, Colomer-Lahiguera S, Spurrier-Bernard G, Latifyan S, Addeo A, Michielin O, Eicher M. Acceptability of an Electronic Patient-Reported Outcomes-Based Model of Care to Monitor Symptoms Related to Cancer Treatment with Immune Checkpoint Inhibitors: Results from the IePRO Randomized Controlled Trial. Semin Oncol Nurs. 2025 Aug;41(4):151903. doi: 10.1016/j.soncn.2025.151903. Epub 2025 May 24. PMID 40413059
- [Derived] da Silva Lopes AM, Colomer-Lahiguera S, Darnac C, Giacomini S, Bugeia S, Gutknecht G, Spurrier-Bernard G, Cuendet M, Muet F, Aedo-Lopez V, Mederos N, Michielin O, Addeo A, Latifyan S, Eicher M. Testing a Model of Care for Patients on Immune Checkpoint Inhibitors Based on Electronic Patient-Reported Outcomes: Protocol for a Randomized Phase II Controlled Trial. JMIR Res Protoc. 2023 Oct 18;12:e48386. doi: 10.2196/48386. PMID 37851498